CLINICAL TRIAL: NCT00004228
Title: Randomized Phase III Study for the Treatment of Newly Diagnosed Disseminated Lymphoblastic Lymphoma or Localized Lymphoblastic Lymphoma
Brief Title: Combination Chemotx in Treating Children or Adolescents With Newly Diagnosed Stg III or Stg IV Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5971; CCG-59701 (Other: Children's Cancer Group); CCG-59701C (Other: Children's Cancer Group); CCG-A5971 (Other: Children's Cancer Group); POG-A5971 (Other: Pediatric Oncology Group); CDR0000067470 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2016-11

CONDITIONS: Lymphoma
Keywords: stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; prednisolone phosphate; Thioguanine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A0 (localized disease Stg I/II) Modified CCG BFM (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Doxorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate
- A1 (Disseminated, No CNS - CCG mod BFM w/out intens (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, doxorubicin hydrochloride, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, prednisone, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate
- A2 (Disseminated, No CNS - CCG mod BFM w/ intens (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, daunorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate
- B2 (CNS+) NHL/BFM-95 w/intens delayed radiation therapy (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, daunorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- B1 (Disseminated CNS- <Amend 7B) NHL/BFM-95 w/out intens (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, doxorubicin hydrochloride, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate
- B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/intens (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, daunorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate
- B1 (Disseminated CNS-) NHL/BFM-95 w/out intens (Experimental): Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, doxorubicin hydrochloride, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate

INTERVENTIONS:
Drug: asparaginase — Given IV
  Other Names: E.coli L-asparaginase; EC 3.5.2.2; colaspase; L-asnase; Elspar; Kidrolase; Crasnitin; Leunase; NSC#109229
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC #26271
Drug: cytarabine — Given IV
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #63878
Drug: daunorubicin hydrochloride — Given IV
  Other Names: daunomycin; rubidomycin; Cerubidine; NSC #82151
Drug: dexamethasone — Given IV
  Other Names: Decadron; Hexadrol; Dexone; Dexameth; NSC #34521
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127
Drug: leucovorin calcium — Given IV
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #003590
  Arms: B1 (Disseminated CNS- <Amend 7B) NHL/BFM-95 w/out intens; B1 (Disseminated CNS-) NHL/BFM-95 w/out intens; B2 (CNS+) NHL/BFM-95 w/intens delayed radiation therapy; B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/intens
Drug: mercaptopurine — Given IV
  Other Names: 6-MP; Purinethol; 6-mercaptopurine; NSC #000755
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; Trexall; NSC #000740
Drug: prednisone — Given IV
  Other Names: Deltasone; Meticorten; Orasone; Liquid Pred; Pediapred; Sterapred; NSC #010023
Drug: thioguanine — Given PO
  Other Names: 6-thioguanine; 2-amino-1,7-dihydro-6H-purine-6-thione; WR-1141; Tabloid; Lanvis; NSC # 751
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; VCR; LCR; NSC #67574
Radiation: radiation therapy
  Arms: B2 (CNS+) NHL/BFM-95 w/intens delayed radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which regimen of combination chemotherapy is most effective for lymphoblastic lymphoma.

PURPOSE: This randomized phase III trial is studying different regimens of combination chemotherapy to compare how well they work in treating children or adolescents with newly diagnosed stage III or stage IV lymphoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival and overall survival of children or adolescents with newly diagnosed disseminated stage III or IV lymphoblastic lymphoma treated with 4 chemotherapy regimens*.
* Determine whether treatment with a regimen without methotrexate maintains the same disease-free survival as NHL/BFM 90 in these patients.
* Determine whether intensification with anthracycline and cyclophosphamide improves disease-free survival in these patients.
* Collect outcome data on uniformly treated patients with localized disease or CNS-positive disease.
* Determine whether rapid reduction in tumor volume by chest radiography and CT scan is predictive of improved outcome in patients treated with these regimens.
* Determine the prevalence of bone marrow involvement at presentation in these patients.
* Determine whether peripheral blood can replace bone marrow in the initial staging of these patients.
* Determine the clinical significance of bone marrow and peripheral blood involvement in these patients.

NOTE: *All patients as of 4/2006 receive treatment on Arm III regimen only

OUTLINE: Patients are stratified by disease characteristics (disseminated lymphoblastic lymphoma vs localized lymphoblastic lymphoma [localized lymphoblastic lymphoma is closed to accrual as of 10/2005]) and age. Patients with CNS negative disseminated lymphoblastic lymphoma are randomized to 1 of 4 treatment arms*. Patients with testicular involvement at diagnosis are nonrandomly assigned to arm IV and do not receive testicular radiotherapy. Patients with localized lymphoblastic lymphoma (closed to accrual as of 10/2005) are not randomized.

NOTE: *All patients as of 4/2006 receive treatment on Arm III only

* Localized lymphoblastic lymphoma (closed to accrual as of 10/2005):

  * Induction (5 weeks): Patients receive vincristine IV and daunorubicin IV over 15 minutes to 2 hours on days 0, 7, 14, and 21; oral prednisone on days 0-27; and asparaginase intramuscularly (IM) on days 3, 5, and 7 and then 3 times a week for 9 doses (during days 8-21). Patients also receive methotrexate intrathecally (IT) on days 7 and 28 and cytarabine IT on day 0.
  * Consolidation (5 weeks): Patients receive methotrexate IT on days 0, 7, 14, and 21 followed by cyclophosphamide IV over 1 hour on days 0 and 14; cytarabine IV on days 0-3, 7-10, 14-17, and 21-24; oral mercaptopurine on days 0-27; and oral prednisone over 10 days.
  * Interim maintenance (8 weeks): Patients receive methotrexate IT on days 0 and 28; oral mercaptopurine on days 0-41; and oral methotrexate on days 7, 14, 21, and 35.
  * Delayed intensification (7 weeks): Patients receive vincristine IV and doxorubicin IV over 15 minutes to 2 hours on days 0, 7, and 14; asparaginase IM on day 3 and then 3 times a week for 6 doses; oral dexamethasone on days 0-30; cyclophosphamide IV over 1 hour on day 28; and cytarabine IV or SC on days 28-31 and 35-38. Patients also receive oral thioguanine on days 28-41 and methotrexate IT on days 28 and 35.
  * Maintenance (84 day course): Patients receive vincristine IV on days 0, 28, and 56; oral prednisone on days 0-4, 28-32, and 56-60; oral methotrexate on days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, and 77; oral mercaptopurine on days 0-83; and methotrexate IT on day 0.
* Disseminated lymphoblastic lymphoma:

  * Arm I (closed to accrual as of 4/2006): Patients receive same induction, consolidation, and interim maintenance therapy schedule as localized lymphoblastic lymphoma patients.

    * Delayed intensification (7 weeks): Patients receive vincristine IV and doxorubicin IV over 15 minutes to 2 hours on days 0, 7, 14, and 21; asparaginase IM on day 3 and then 3 times a week for 6 doses; and oral dexamethasone on days 0-28. Patients also receive cyclophosphamide IV over 1 hour on day 35; cytarabine IV or SC on days 35-38 and 42-45; oral thioguanine on days 35-48; and methotrexate IT on days 35 and 42.
    * Maintenance (84 day course): Patients receive same therapy as localized lymphoblastic lymphoma patients, except methotrexate IT is administered on day 0 and 28 (for first 4 courses).
  * Arm II (closed to accrual as of 4/2006): Patients receive consolidation, interim maintenance, and maintenance therapy as in arm I.

    * Induction (5 weeks): Patients receive vincristine IV on days 0, 7, 14, and 21; daunorubicin IV over 48 hours on days 0-2; oral prednisone on days 0-27; and asparaginase IM on days 3, 5, and 7 and then 3 times a week for 9 doses (during days 8-21). Patients also receive methotrexate IT on days 7 and 28; cyclophosphamide IV over 1 hour on day 2; and cytarabine IT on day 0.
    * Delayed intensification (7 weeks): Patients receive vincristine IV on days 0, 7, 14, 21; daunorubicin IV over 48 hours on days 0-2; asparaginase IM on day 3 and then 3 times a week for 6 doses; and oral dexamethasone on days 0-28. Patients also receive cyclophosphamide IV over 1 hour on days 2 and 35; cytarabine IV or SC on days 35-38 and 42-45; oral thioguanine on days 35-48; and methotrexate IT on days 35 and 42.
  * Arm III:

    * Induction (5 weeks): Patients receive vincristine IV and daunorubicin IV over 1 hour on days 0, 7, 14, and 21 and oral prednisone on days 0-37. Patients also receive asparaginase IM on day 11 and then 3 times a week for 9 doses; methotrexate IT on days 7 and 28; and cytarabine IT on day 0.
    * Consolidation (5 weeks): Patients receive methotrexate IT and cyclophosphamide IV over 1 hour on days 0 and 14; cytarabine IV or SC on days 0-3, 7-10, 14-17, and 21-24; oral mercaptopurine on days 0-27; and oral prednisone over 10 days.
    * Interim maintenance (9 weeks): Patients receive methotrexate IT and IV on days 7, 21, 35, and 49; oral mercaptopurine on days 0-55; and leucovorin calcium IV at 42, 48, and 54 hours after methotrexate IV.
    * Delayed intensification (10 weeks): Patients receive vincristine IV and doxorubicin IV over 1 hour on days 0, 7, 14, and 21; asparaginase IM on day 3 and then 3 times a week for 6 doses; and oral dexamethasone on days 0-29. Patients also receive cyclophosphamide IV over 1 hour on day 35; cytarabine IV on days 35-38 and 42-45; oral thioguanine on days 35-48; and methotrexate IT on days 35 and 42.
    * Maintenance (84 day courses): Patients receive vincristine IV on days 0, 28, and 56; oral prednisone on days 0-4, 28-32, and 56-60; oral methotrexate on days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, and 77; and oral mercaptopurine on days 0-83.
  * Arm IV (closed to accrual as of 4/2006): Patients receive consolidation and interim maintenance therapy as in arm III.

    * Induction: Patients receive vincristine IV on days 0, 7, 14, and 21; daunorubicin IV over 48 hours on days 0-2; oral prednisone on days 0-37; asparaginase IM on day 11 and then 3 times a week for 9 doses; methotrexate IT on days 7, 14, 21, and 28; cyclophosphamide IV on day 2; and cytarabine IT on day 0.
    * Delayed intensification (10 weeks): Patients receive vincristine IV on days 7, 14, 21, and 28; daunorubicin IV over 48 hours on days 0-2; asparaginase IM on day 3 and then 3 times a week for 6 doses; and oral dexamethasone on days 0-29. Patients also receive cyclophosphamide IV over 1 hour on days 2 and 35; cytarabine IV on days 35-38 and 42-45; oral thioguanine on days 35-48; and methotrexate IT on days 35 and 42.
    * Maintenance (84 day courses): Patients receive therapy as in arm III. Patients who are over 1 year of age and have CNS disease at diagnosis undergo cranial radiotherapy once daily 5 days a week beginning on day 0. Patients over 2 years of age undergo radiotherapy over 11-14 days (6-9 days for 1-2 years of age).

Patients are followed monthly for one year, every 3 months for 1 year, every 6 months for 1.5 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 250-400 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed disseminated lymphoblastic lymphoma or localized lymphoblastic lymphoma*

  * Less than 25% tumor cells in the bone marrow
  * Previously untreated (prior intrathecal cytarabine allowed if protocol therapy begins within 72 hours)
  * Stage III or IV disease
* NOTE: *Localized lymphoblastic lymphoma is closed to accrual as of 10/2005

PATIENT CHARACTERISTICS:

Age:

* 1 to 30

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* Adequate cardiac function

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Emergency steroid therapy (if required) must be started within 72 hours prior to protocol therapy

Radiotherapy:

* Emergency radiotherapy (if required) must be started within 72 hours prior to protocol therapy

Surgery:

* Not specified

Other:

* No other prior therapy except for emergency treatment of airway obstruction and/or superior vena cava syndrome

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 393 (Actual)
Dates: Start 2000-06; Primary Completion 2008-08 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minnie Abromowitch, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (176):
- United States (152):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Scarborough, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Australia (5):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Royal Children's Hospital, Herston, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Patel JL, Smith LM, Anderson J, Abromowitch M, Campana D, Jacobsen J, Lones MA, Gross TG, Cairo MS, Perkins SL. The immunophenotype of T-lymphoblastic lymphoma in children and adolescents: a Children's Oncology Group report. Br J Haematol. 2012 Nov;159(4):454-61. doi: 10.1111/bjh.12042. Epub 2012 Sep 21. PMID 22994934
- [Result] Termuhlen AM, Smith LM, Perkins SL, Lones M, Finlay JL, Weinstein H, Gross TG, Abromowitch M. Outcome of newly diagnosed children and adolescents with localized lymphoblastic lymphoma treated on Children's Oncology Group trial A5971: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2012 Dec 15;59(7):1229-33. doi: 10.1002/pbc.24149. Epub 2012 Apr 5. PMID 22488718
- [Result] Coustan-Smith E, Sandlund JT, Perkins SL, Chen H, Chang M, Abromowitch M, Campana D. Minimal disseminated disease in childhood T-cell lymphoblastic lymphoma: a report from the children's oncology group. J Clin Oncol. 2009 Jul 20;27(21):3533-9. doi: 10.1200/JCO.2008.21.1318. Epub 2009 Jun 22. PMID 19546402
- [Result] Abromowitch M, Termuhlen A, Chang M, et al.: High-dose methotrexate and early intensification of therapy do not improve 3 year EFS in children and adolescents with disseminated lymphoblastic lymphoma: results of the randomized arms of COG A5971. [Abstract] Blood 112 (11): A-3610, 2008.
- [Result] Smock KJ, Nelson M, Tripp SR, Sanger WG, Abromowitch M, Cairo MS, Perkins SL; Children's Oncology Group. Characterization of childhood precursor T-lymphoblastic lymphoma by immunophenotyping and fluorescent in situ hybridization: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2008 Oct;51(4):489-94. doi: 10.1002/pbc.21666. PMID 18618503
- [Result] Coustan-Smith E, Abromowitz M, Sandlund JT, et al.: A novel approach for minimal residual disease detection in childhood T-cell lymphoblastic lymphoma (T-LL): a Children's Oncology Group report. [Abstract] Blood 110 (11): A-3564, 2007.

RESULTS

PARTICIPANT FLOW:
Groups:
- B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment: Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, doxorubicin hydrochloride, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
Period: Overall Study
Arm/Group | A0 (Localized Disease Stg I/II) Modified CCG BFM | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens | A2 (Disseminated, No CNS - CCG Mod BFM w/ Intens | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment
Started | 60 | 66 | 65 | 13 | 67 | 65 | 57
Completed | 51 | 51 | 46 | 6 | 51 | 51 | 45
Not Completed | 9 | 15 | 19 | 7 | 16 | 14 | 12
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 6 | 5 | 3 | 9 | 8 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 3 | 2 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 5 | 2 | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0 | 2 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — ineligible | 4 | 2 | 4 | 1 | 1 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- A2 (Disseminated, No CNS - CCG Mod BFM w/Intens: Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, daunorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
- Total: Total of all reporting groups
Arm/Group | A0 (Localized Disease Stg I/II) Modified CCG BFM | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens | A2 (Disseminated, No CNS - CCG Mod BFM w/Intens | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment | Total
Number analyzed (Participants) | 60 | 66 | 65 | 13 | 67 | 65 | 57 | 393
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 62 | 63 | 12 | 65 | 62 | 52 | 373
  Between 18 and 65 years | 3 | 4 | 2 | 1 | 2 | 3 | 5 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.9) | 10.5 (5.2) | 10 (4.8) | 11.4 (5.3) | 10.2 (5.1) | 10.6 (5.1) | 11.5 (5.1) | 10.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 9 | 4 | 20 | 16 | 17 | 108
  Male | 37 | 47 | 56 | 9 | 47 | 49 | 40 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 4 | 3 | 9 | 12 | 3 | 55
  Not Hispanic or Latino | 47 | 53 | 58 | 10 | 58 | 47 | 52 | 325
  Unknown or Not Reported | 2 | 0 | 3 | 0 | 0 | 6 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 3 | 0 | 3 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 3 | 5 | 9 | 2 | 6 | 5 | 11 | 41
  White | 53 | 56 | 48 | 10 | 54 | 53 | 41 | 315
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 02 | 2
  Unknown or Not Reported | 3 | 2 | 4 | 1 | 4 | 7 | 2 | 23
Region of Enrollment [Number; unit: participants]
  United States | 48 | 58 | 57 | 12 | 62 | 58 | 51 | 346
  Canada | 5 | 3 | 6 | 1 | 4 | 4 | 4 | 27
  Australia | 7 | 4 | 1 | 0 | 0 | 3 | 1 | 16
  Switzerland | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Assessed by time to treatment failure, occurrence of second malignant neoplasm, or death from any cause. Statistical analysis will be to estimate the difference in the proportion of patients treated with each therapy who are long-term event-free survivors due either to the difference between the backbone therapy regimens (CCG BFM vs NHL/BFM-95), or due to the intensification.
Time Frame: 5 years
Population: There were 19 total ineligible patients, 4 for A0, 2 for A1, 4 for A2, 1 for B2 (CNS+), 1 for B2 (Disseminated), 2 for B1 (CNS-), and 5 for B1 (NHL additional enrollment) not included in outcome measure analysis.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | A0 (Localized Disease Stg I/II) Modified CCG BFM | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens | A2 (Disseminated, No CNS - CCG Mod BFM w/ Intens | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment
Number analyzed (Participants) | 56 | 64 | 61 | 12 | 66 | 63 | 52
percentage of particpants | 88 [76 to 95] | 82 [70 to 90] | 80 [67 to 89] | 63 [29 to 85] | 82 [70 to 89] | 84 [72 to 91] | 90 [78 to 96]
Statistical Analysis 1: Comparison: A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens vs A2 (Disseminated, No CNS - CCG Mod BFM w/ Intens vs B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy vs B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens vs B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment; A Cox model was used to assess evidence of a difference in event-free survival comparing regimens A1+A2 ("A: CCG BFM") to regimens B1+B2 ("B: NHL/BFM-95") while adjusting for the other intervention through stratification; Test type: Superiority or Other; p = .97, Regression, Cox
Statistical Analysis 2: Comparison: A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens vs A2 (Disseminated, No CNS - CCG Mod BFM w/ Intens vs B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy vs B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens; A Cox model was used to assess evidence of a difference in event-free survival comparing A1+B1 ("1: no intensification") to A2 +B2 ("2: intensification"), while adjusting for the other intervention through stratification; Test type: Superiority or Other; p = .63, Regression, Cox

2. Secondary Outcome: Percentage of Patients With Overall Survival as Assessed by Time to Death
Description: Overall survival will be computed by measuring the rate of deaths during induction due primarily to treatment toxicity and cumulative incidence of toxic deaths in induction or deaths in remission overall and separately for treatment groups defined by the two design factors.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A0 (Localized Disease Stg I/II) Modified CCG BFM | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens | A2 (Disseminated, No CNS - CCG Mod BFM w/Intens | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment
Number analyzed (Participants) | 56 | 64 | 61 | 12 | 66 | 63 | 52
percentage of participants | 96 [84 to 99] | 84 [72 to 91] | 88 [76 to 94] | 81 [42 to 95] | 85 [73 to 91] | 85 [74 to 92] | 92 [80 to 97]

ADVERSE EVENTS:
Description: There were 19 total ineligible patients, 4 for A0, 2 for A1, 4 for A2, 1 for B2 (CNS+), 1 for B2 (Disseminated), 2 for B1 (CNS-), and 5 for B1 (NHL additional enrollment). All ineligible patients excluded from adverse event reporting.
Groups:
- B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens; B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment: Phase I - 5 week induction (Vincristine Sulfate, daunorubicin hydrochloride, Cyclophosphamide, L-Asparaginase, Intrathecal Cytarabine, Intrathecal Methotrexate, Prednisone). Phase II - 5 week consolidation (Mercaptopurine, Cyclophosphamide, Cytarabine, Intrathecal Methotrexate, Prednisone). Phase III - 8 week Interim Maintenance (Mercaptopurine, Methotrexate, Intrathecal Methotrexate, Leucovorin Calcium). Phase IV - 7 week Delayed Intensification (Vincristine Sulfate, Cyclophosphamide, daunorubicin, L-Asparaginase, Dexamethasone, Cyclophosphamide, Thioguanine, Cytarabine, Intrathecal Methotrexate). Phase V - 12 week courses (Vincristine Sulfate, Prednisone, Mercaptopurine, Methotrexate, Intrathecal Methotrexate)
Arm/Group | A0 (Localized Disease Stg I/II) Modified CCG BFM | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens | A2 (Disseminated, No CNS - CCG Mod BFM w/Intens | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment
Serious Adverse Events (participants affected / at risk) | 8/56 | 8/64 | 13/61 | 0/12 | 12/66 | 9/63 | 1/52
Other Adverse Events (participants affected / at risk) | 56/56 | 64/64 | 60/61 | 10/12 | 66/66 | 62/63 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A0 (Localized Disease Stg I/II) Modified CCG BFM (N=56) | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens (N=64) | A2 (Disseminated, No CNS - CCG Mod BFM w/Intens (N=61) | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy (N=12) | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens (N=66) | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens (N=63) | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment (N=52)
Bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular/Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular/General-Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter-related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cortical blindness, Anxiety, agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fever, Increase BP, Back pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache, Vomiting, Nausea, Pancytopenia, Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 3 (4) | 4 (5) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection/Febrile Neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection/Febrile Neutropenia (sepsis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (8) | 5 (5) | 7 (7) | 0 (0) | 12 (16) | 7 (10) | 0 (0)
Lt Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
N/V, Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial thromboplastin time (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelets (Investigations) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
SGOT (AST) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
SGPT (ALT) (Investigations) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (4) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clot (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
difficulty with speech, Left sided numbness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A0 (Localized Disease Stg I/II) Modified CCG BFM (N=56) | A1 (Disseminated, No CNS - CCG Mod BFM w/Out Intens (N=64) | A2 (Disseminated, No CNS - CCG Mod BFM w/Intens (N=61) | B2 (CNS+) NHL/BFM-95 w/Intens Delayed Radiation Therapy (N=12) | B2 (Disseminated,CNS- (< Amend 7B)) NHL/BFM-95 w/Intens (N=66) | B1 (Disseminated CNS-) NHL/BFM-95 w/Out Intens (N=63) | B1 (NHL/BFM-95 w/Out Intens) Additional Enrollment (N=52)
Allergic reaction/hypersensitivity (Immune system disorders) | 1 (2) | 4 (5) | 1 (1) | 1 (1) | 3 (4) | 3 (3) | 1 (1)
Autoimmune reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergy/Immunology (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inner ear/hearing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear/hearing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Auditory/Hearing (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 56 (509) | 64 (533) | 60 (520) | 10 (69) | 66 (530) | 62 (496) | 52 (476)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Investigations) | 56 (532) | 64 (552) | 60 (536) | 10 (72) | 66 (556) | 62 (505) | 52 (476)
Lymphopenia (Investigations) | 12 (40) | 13 (52) | 10 (40) | 1 (5) | 15 (39) | 8 (26) | 9 (29)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 28 (86) | 45 (139) | 40 (116) | 5 (14) | 36 (114) | 37 (98) | 27 (79)
Platelets (Investigations) | 56 (469) | 64 (523) | 60 (499) | 10 (69) | 66 (520) | 61 (468) | 52 (476)
Transfusion: Platelets (Blood and lymphatic system disorders) | 19 (28) | 14 (24) | 18 (21) | 3 (5) | 14 (22) | 12 (15) | 9 (12)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 24 (40) | 29 (54) | 25 (42) | 3 (7) | 30 (51) | 27 (45) | 28 (30)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Vasovagal episode (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular/Arrhythmia (Cardiac disorders) | 48 (406) | 59 (469) | 56 (458) | 10 (63) | 60 (475) | 60 (427) | 52 (476)
Cardiac left ventricular function (Cardiac disorders) | 52 (428) | 61 (482) | 56 (462) | 10 (62) | 61 (482) | 61 (436) | 52 (476)
Edema (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 4 (4) | 6 (7) | 0 (0) | 7 (7) | 5 (5) | 9 (11)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Pericardial effusion/pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombosis/embolism (Vascular disorders) | 2 (2) | 7 (7) | 4 (4) | 0 (0) | 6 (6) | 5 (7) | 6 (6)
Cardiovascular/General (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrinogen (Investigations) | 3 (4) | 3 (3) | 4 (4) | 0 (0) | 6 (6) | 7 (7) | 4 (5)
Partial thromboplastin time (PTT) (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 2 (4) | 0 (0)
Prothrombin time (PT) (Investigations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 0 (0)
Coagulation (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3 (6) | 3 (7) | 4 (5) | 2 (2) | 5 (7) | 1 (2) | 2 (2)
Fever (General disorders) | 5 (7) | 2 (3) | 5 (7) | 0 (0) | 6 (8) | 12 (16) | 4 (4)
Rigors, chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (General disorders) | 1 (2) | 5 (14) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight loss (General disorders) | 0 (0) | 2 (4) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Constitutional Symptoms (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (8) | 1 (1) | 0 (0) | 3 (9) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6) | 4 (6) | 1 (2) | 5 (11) | 5 (5) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound-infectious (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Wound-non infectious (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 7 (10) | 0 (0) | 1 (1) | 2 (4) | 2 (2)
Cushingoid appearance (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 2 (4) | 1 (1) | 1 (1)
SIADH (syndrome of inappropriate antidiuretic hormone) (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Endocrine (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 5 (9) | 0 (0) | 7 (12) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 7 (13) | 5 (7) | 0 (0) | 8 (9) | 7 (9) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 4 (4) | 0 (0) | 7 (10) | 8 (10) | 3 (8)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 7 (7) | 7 (13) | 7 (9) | 0 (0) | 4 (6) | 9 (11) | 3 (4)
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (5) | 2 (3)
Fistula-intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula-rectal/anal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Mouth dryness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (8) | 9 (16) | 5 (14) | 1 (1) | 9 (14) | 8 (11) | 8 (10)
Pancreatitis (Gastrointestinal disorders) | 52 (431) | 61 (481) | 56 (458) | 10 (62) | 63 (481) | 61 (436) | 52 (476)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 4 (7) | 9 (13) | 7 (11) | 2 (2) | 17 (21) | 20 (24) | 15 (19)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12) | 7 (15) | 8 (11) | 1 (1) | 11 (18) | 12 (17) | 6 (9)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CNS hemorrhage/bleeding (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 4 (11) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 3 (5) | 2 (2)
Bilirubin (Investigations) | 53 (444) | 61 (492) | 57 (483) | 10 (63) | 65 (505) | 62 (454) | 52 (476)
GGT (Investigations) | 1 (3) | 3 (9) | 3 (3) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Hepatic enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (12) | 5 (9) | 7 (9) | 0 (0) | 6 (7) | 4 (5) | 4 (4)
SGOT (AST) (Investigations) | 54 (469) | 62 (502) | 59 (492) | 10 (63) | 65 (509) | 62 (468) | 52 (476)
SGPT (ALT) (Investigations) | 54 (487) | 63 (516) | 59 (505) | 10 (67) | 65 (520) | 62 (482) | 52 (476)
Hepatic (Hepatobiliary disorders) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter-related infection (Infections and infestations) | 51 (430) | 63 (483) | 58 (460) | 10 (62) | 63 (481) | 62 (443) | 52 (476)
Febrile neutropenia (Blood and lymphatic system disorders) | 56 (451) | 62 (490) | 59 (472) | 10 (66) | 64 (486) | 62 (446) | 52 (476)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 54 (441) | 63 (488) | 59 (469) | 10 (64) | 64 (488) | 62 (440) | 52 (476)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 53 (438) | 63 (485) | 57 (461) | 10 (62) | 63 (488) | 61 (445) | 52 (476)
Infection/Febrile Neutropenia (Infections and infestations) | 50 (410) | 58 (467) | 58 (460) | 10 (65) | 60 (473) | 60 (425) | 52 (476)
Lymphatics (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Amylase (Investigations) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 4 (6) | 0 (0)
Bicarbonate (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (6) | 1 (1)
Hypercholesterolemia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (15) | 13 (27) | 13 (25) | 2 (3) | 13 (20) | 16 (30) | 14 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 2 (2) | 1 (1) | 6 (8) | 2 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 1 (2) | 4 (7) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 5 (6) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (11) | 7 (9) | 10 (17) | 2 (2) | 13 (13) | 9 (12) | 9 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 4 (4) | 1 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 10 (19) | 8 (15) | 11 (20) | 0 (0) | 10 (11) | 13 (15) | 19 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 5 (6) | 2 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (10) | 5 (6) | 7 (10) | 1 (1) | 13 (15) | 10 (13) | 20 (26)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8) | 5 (6) | 4 (6) | 0 (0) | 7 (7) | 6 (6) | 4 (4)
Lipase (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Metabolic/Laboratory (Investigations) | 3 (7) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (4) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 52 (430) | 61 (480) | 57 (460) | 10 (62) | 61 (477) | 61 (435) | 52 (476)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 51 (428) | 61 (482) | 56 (456) | 10 (62) | 61 (478) | 61 (435) | 52 (476)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Delusions (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness/lightheadedness (Nervous system disorders) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Leukoencephalopathy associated radiological findings (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Memory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mood alteration-depression (Psychiatric disorders) | 0 (0) | 4 (9) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neuropathy - cranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neuropathy - motor (Nervous system disorders) | 3 (3) | 4 (5) | 7 (7) | 0 (0) | 9 (11) | 5 (5) | 3 (3)
Neuropathy - sensory (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 6 (7) | 5 (7) | 4 (5)
Personality/behavioral (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Seizure(s) (Nervous system disorders) | 51 (432) | 62 (481) | 56 (456) | 10 (62) | 63 (481) | 61 (437) | 52 (476)
Speech impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurology (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tearing (watery eyes) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision-photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (5) | 6 (10) | 7 (8) | 1 (1) | 13 (13) | 4 (5) | 4 (4)
Arthralgia (joint pain) (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Bone pain (General disorders) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Earache (otalgia) (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Headache (General disorders) | 3 (6) | 9 (23) | 9 (10) | 3 (5) | 5 (11) | 5 (7) | 5 (5)
Myalgia (muscle pain) (General disorders) | 2 (2) | 5 (8) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Neuropathic pain (General disorders) | 1 (2) | 5 (8) | 5 (6) | 2 (3) | 7 (7) | 7 (11) | 2 (2)
Pelvic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleuritic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rectal or perirectal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 6 (7) | 5 (7) | 1 (1) | 8 (11) | 9 (11) | 5 (7)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 5 (8) | 2 (2) | 1 (1) | 2 (5) | 7 (9) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 4 (4) | 4 (4) | 2 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (3) | 2 (2) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice changes/stridor/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Serum Creatinine (Investigations) | 51 (438) | 62 (482) | 57 (467) | 10 (62) | 63 (492) | 61 (450) | 52 (476)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 51 (431) | 61 (480) | 57 (457) | 10 (62) | 63 (480) | 61 (436) | 52 (476)
Urinary electrolyte wasting (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Secondary malignancy - Other (Specify type, excludes metastastic tumors) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irregular menses (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syndromes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (9) | 3 (5) | 2 (4) | 1 (2) | 6 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.